CLINICAL TRIAL: NCT04497649
Title: Sofosbuvir Containing Regimens in Treatment of COVID 19 Patients: A Randomized Controlled Trial.
Brief Title: Sofosbuvir Containing Regimens in Treatment of COVID 19 Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tanta sofosbuvir covid
Record Dates: First submitted 2020-08-01; First posted 2020-08-04 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Sofosbuvir; daclatasvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sofosbuvir and Daklatasuvir (Experimental): Sofosbuvir and Daklatasuvir with standard of care treatment
  Interventions: Drug: Sofosbuvir; Drug: Daclatasvir
- Standard of care treatment (No Intervention): Standard of care treatment

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir once daily
  Other Names: Mpiviropack, Sovaldy, soflanork
  Arms: Sofosbuvir and Daklatasuvir
Drug: Daclatasvir — daclatasuvir once daily
  Other Names: daklinza, daklanork
  Arms: Sofosbuvir and Daklatasuvir

SUMMARY:
efficacy and safety of Sofosbuvir containing regimens in treatment of COVID-19 Egyptian patients,

DETAILED DESCRIPTION:
The study aims to assess Sofosbuvir containing regimens in treatment of COVID-19 Egyptian patients,

ELIGIBILITY:
Inclusion Criteria:

* COVID 19 positive patients

Exclusion Criteria:

* COVID-19 patients with critical manifestations.
* Sepsis.
* Acute respiratory distress syndrome (ARDS).
* Decompensated liver disease (Child-Pugh class B or C disease).
* Chronic renal impairment.
* Patients with blood diseases (severe anemia, thalassemia, ITP, leukemia ….).
* Ischemic heart disease within the last 6 months.
* Chronic pulmonary disease.
* Malignancy.
* Pregnancy or breastfeeding.
* Hypersensitivity to sofosbuvir or ribavirin.
* Patients with organ transplant.
* Unwilling to participate in our study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with improvement or mortality | 1 month
  The number of patients with improvement or mortality

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Salama, Lecturer, Principal Investigator — Tanta University - Faculty of Medicine; sherief Abd-Elsalam, ass. Prof., Principal Investigator — Tanta University Faculty of medicine; Ahmed Cordie, lecturer, Principal Investigator — Cairo University; Gamal Esmat, Professor, Principal Investigator — Cairo University
Locations (1):
- Cairo and Tanta Universitities, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No